CLINICAL TRIAL: NCT05764941
Title: Real World Study of Inetetamab Combined With Pyrotinib and Vinorelbine as First-line to Third-line Treatment for Trastuzumab Resistant HER2-positive Metastatic Breast Cancer: a Multicenter, Retrospective Study
Brief Title: Inetetamab Combined With Pyrotinib and Vinorelbine as First-line to Third-line Treatment for HER2-positive Metastatic Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ILLUMINE
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Vinorelbine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: Patients receive initetamab combined with pyrotinib and vinorelbine after trastuzumab progression.
  Interventions: Drug: Inetetamab; Drug: Pyrotinib; Drug: Vinorelbine

INTERVENTIONS:
Drug: Inetetamab — 8mg/kg for the first dose, 6mg/kg for the following doses, every 3 weeks for one cycle.
Drug: Pyrotinib — 400mg, oral, every day.
Drug: Vinorelbine — 25 mg/m2, D1, D8, every 3 weeks for one cycle.

SUMMARY:
This is a real world study to evaluate the efficacy and safety of inetetamb combined with pyrotinib and vinorelbine as first-line to third-line treatment after trastuzumab progression in HER2-positive metastatic breast cancer.

DETAILED DESCRIPTION:
HER2-positive breast cancers account for 15%-20% of all breast cancers. Despite trastuzumab has significantly improved the survival of patients with HER2-positivie metastatic breast cancer as the first-line standard treatment, the selection of drugs after trastuzumab treatment failure remains difficulty and challenge. Inetetamab, a new antibody to optimize the ADCC effect, has shown great effectiveness in treating HER2-positive metastatic breast cancer, but therapies subsequent to trastuzumab progression are still controversial. Pyrotinib, another second-line HER2 targeted drug, is a typical representative of TKI drugs, which not only has a strong HER2 antagonistic effect but also can synergize with monoclonal antibodies to amplify the ADCC effect. Here, investigators studied the efficacy and safety of inetetamb combined with pyrotinib and vinorelbine as first-line to third-line treatment after trastuzumab progression, so as to provide new ideas for the treatment of patients with HER2-positive metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female and 18-80 years old;
2. The patient was diagnosed as HER2-positive breast cancer by histopathology (HER2 positive (IHC +++ or IHC++ but FISH/CISH+ ));
3. All patients have previously received ≤ 2 lines chemotherapy for metastatic breast cancer;
4. Patients received inetetamab combined with pyrotinib and vinorelbine after trastuzumab failure;
5. According to RECIST 1.1, patients with at least one target lesion or simple bone metastasis can be evaluated;
6. ECOG score of physical status was less than 2, and the expected survival time was not less than 3 months;
7. Complete and traceable medical data.

Exclusion Criteria:

1. Incomplete medical data;
2. The investigator believes that the patient is not suitable to enter this study.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HER2-positive metastatic breast cancer patients received inetetamab combined with pyrotinib and vinorelbine after trastuzumab failure
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 years
  Progression-free survival estimated using Kaplan-Meier methods is defined as the time from the date of informed consent to the earlier of death or disease progression. Patients alive without disease progression are censored at the date of last disease evaluation. Progressive disease (PD) based on RECIST 1.1 is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. Equivocal progression of non-target lesions also qualifies as PD.
Objective Response Rate (ORR) | 2 years
  The overall response rate is defined as the percentage of patients with a best overall response of CR or PR relative to the appropriate analysis set

SECONDARY OUTCOMES:
The Number of Participants Who Experienced Adverse Events (AE) | 2 years
  Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). AE grade were defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events).

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No